CLINICAL TRIAL: NCT05079139
Title: Musset's Surgical Technique: Evaluation of Long-term Results (LONGOMUSSET)
Acronym: LONGOMUSSET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LONGOMUSSET
Record Dates: First submitted 2021-10-05; First posted 2021-10-15 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Rectovaginal Fistula; Obstetric Complication
Keywords: surgical technique of Musset
MeSH Terms: conditions — Rectovaginal Fistula

STUDY DESIGN:
Intervention Model Description: Descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgical technique of Musset (Other)
  Interventions: Procedure: surgical technique of Musset

INTERVENTIONS:
Procedure: surgical technique of Musset — The one-stage rectovaginal fistula cure according to Musset is an intervention indicated in the treatment of simple post-obstetrical or simple post-surgical rectovaginal fistulas.
  The procedure consists in performing a perineal section to the perineal section to the fistula pathway in order to perform local excision followed by a repair plane by plane with rectal and anal closure, then of the external sphincter of the anus, and interposition of the deep and superficial transverse elevator and perineal muscles before closing the vagina and perineum.

SUMMARY:
The surgical technique of Musset has shown its effectiveness for the cure of recto-vaginal fistulas. Recto-vaginal fistulas are mostly post-obstetric (88%).

The objective of this study is to investigate the outcome of patients who underwent a Musset surgical technique, as well as their postoperative functional and anatomical results at a distance from the procedure.

DETAILED DESCRIPTION:
Obstetric fistulas affect more than 2 million women worldwide with 50,000 to 100,000 cases per year and are responsible for symptoms that can alter the quality of life.

Among fistulas, recto-vaginal fistulas are responsible for disabling symptoms such as the emission of gas and/or stool through the vagina, local infections with purulent and/or malodorous discharge from the vagina, and even dyspareunia. These disabling symptoms constitute a real psycho-social burden for the patients who suffer from them as demonstrated in the study of Singh et al. carried out in India where up to 79.5% felt socially isolated. In developing countries, women with fistula are often abandoned by their husbands and rejected by their families and communities.

Recto-vaginal fistulas are mostly post-obstetric (88%). Indeed, in a study by Goldaber et al. of 24,000 vaginal births, an incidence of 1.7% of grade 4 tears and 0.5% of recto-vaginal fistulas was noted. However, recto-vaginal fistulas can be related to other causes: local infection, post-traumatic (violence, surgery), chronic inflammatory bowel disease (Crohn's ++), radiotherapy, carcinoma or congenital.

The surgical technique of Musset, initially described in 1963, has shown its effectiveness for the cure of recto-vaginal fistulas. In Soriano's retrospective study, 48 patients had undergone recto-vaginal fistula repair using the Musset surgical technique: 25 of the fistulas were of obstetrical origin, 11 of infectious origin, 7 in the context of inflammatory bowel disease and 3 post-surgical. Of the 48 patients, 63% had a history of recto-vaginal fistula treatment, 85% had gas incontinence and 75% had stool incontinence. A total of 47 patients had a satisfactory anatomical and functional outcome with a success rate of 100% for post chronic inflammatory bowel disease fistulas and 98% for patients with a surgical history. Since then, the indication for this procedure has been extended to the treatment of obstetrical perineal sequelae with damage to the external sphincter. In this case, the procedure is usually done in one operation and not two as initially described.

Although this condition affects a significant number of women (mainly in developing countries), few large studies have looked at the results of this technique and the literature is still relatively poor. In particular, no study has looked at the long-term and very long-term results of this surgical technique to definitively demonstrate its benefit, which is all the more fundamental as this pathology essentially affects young women.

The objective of this study is to investigate the outcome of patients who underwent a Musset surgical technique, as well as their postoperative functional and anatomical results at a distance from the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent Musset surgery between January 1, 2002 and December 31, 2020 in the Obstetrics and Reproductive Medicine Department of Intercommunal Hospital Center of Créteil
* Patients who gave their consent to participate in this study
* Patients affiliated with a social security plan

Exclusion Criteria:

* Patients who have undergone rectovaginal fistula treatment using a technique other than the Musset technique
* Patients lost to follow-up
* Patients under legal protection (guardianship, curatorship, safeguard of justice, family habilitation and mandate of future protection activated)

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Presence of gas and/or stool incontinence more than 6 months after surgery | Day 1
  To determine the anatomical and functional results in the long term after cure of recto vaginal fistula according to the Musset technique through questionnaire and auscultation

SECONDARY OUTCOMES:
Questionnaire Short Form 36 (SF 36) (0 to 100) | Day 1
  Assessment of quality of life and overall satisfaction through validated questionnaire
Questionnaire World Health Organization Quality of Life-Bref (WHOQOL-Bref) (0 to 100 in 4 fields) | Day 1
  Assessment of mental health through validated questionnaire
Questionnaire Female Sexual Function Index (FSFI) (2 to 36) | Day 1
  Assessment of sexual quality of life through validated questionnaire
Questionnaire Sexual Activity Questionnaire (SAQ) | Day 1
  Assessment of sexual quality of life through validated questionnaire
Cleveland Score (0 to 20) | Day 1
  Evaluation of the quality of the anatomical restitution through validated questionnaire
Patient Global Impression and Improvement (PGI-I) (1 to 7) | Day 1
  Evaluation of the global impression and improvement to describe as best as possible how your problems are now, compared to how they were compared to what they were before the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No